CLINICAL TRIAL: NCT00342537
Title: Clinical, Genetic, Behavioral, Laboratory and Epidemiologic Studies of Familial Testicular Germ Cell Tumors
Brief Title: Genetics of Familial Testicular Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904076; 04-C-N076; NCT00897598 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Testicular Cancer
Keywords: Pathology; Genetics; Testicular Cancer; Familial; Cancer Epidemiology
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Formalin-fixed, paraffin-imbedded H&E tissue sections from familial and sporadic testicular cancer tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a collaboration between the Clinical Genetics Branch of the National Cancer Institute and the International Testicular Cancer Linkage Consortium (ITCLC). The primary goal of the ITCLC is mapping and cloning susceptibility genes for familial TGCT. The objectives of the current study are to:

* Identify the genes responsible for testicular germ cell tumor (TGCT) (testicular cancer) in families with an inherited tendency to develop the disease
* Determine if the genes which predispose to developing testicular cancer also increase the risk of other specific types of cancer among first- and second-degree relatives of patients with TGCT
* Determine if the microscopic appearance of familial testicular cancers is different from that of non-familial TGCT

Patients and family members recruited by the ITCLC in the United Kingdom, the Netherlands, and Norway are eligible for this study. Individuals with the following medical criteria may participate:

* Patients with testicular germ cell cancer who have at least one other blood relative with the disease
* Family members of patients (first- and second-degree relatives)

Participants undergo the following procedures:

* Fill out questionnaires for providing information about a history of cancer in all blood relatives, including parents, siblings, children, grandparents, aunts, uncles, and cousins, and a history of undescended testes in male blood relatives. Participants may be asked permission to contact family members to request their help in the study as well.
* Provide a blood sample for genetic testing related to TGCT (except in children under 16 years old).
* Review of medical records and examination of tumor specimen (patients with TGCT only).
* Confirmation of the diagnosis of other types of cancer in these same families (medical records, pathology repots)
* Review of the testicular cancer tissue obtained at the time of surgery from members of multiple case families, and comparison of these findings with a series of TGCT which have developed in men without a family history.

DETAILED DESCRIPTION:
Familial clustering of testicular germ cell tumors (TGCT) is well-documented, and a family history of TGCT is associated with an increased risk of this disease. The International Testicular Cancer Linkage Consortium (ITCLC) has assembled 350 multiple case TGCT families in support of a linkage effort that provisionally mapped a susceptibility gene to chromosome Xq27 in a subset of these kindreds. However, familial TGCT is genetically heterogeneous, thus increasing the need for meticulous case definition and classification in ongoing genetic and etiologic studies. The histopathologic classification of TGCT is very complicated; few pathologists have extensive experience reviewing this uncommon tumor. Basing epidemiologic studies upon local pathology reports may result in failure to recognize etiologically critical TGCT subsets of the kind which have been central to suspecting and defining various hereditary cancer syndromes, such as the multiple inherited renal cancer disorders.

Few studies have addressed the risk of cancer among relatives of sporadic TGCT patients. Recent reports suggest a 20% increase in overall cancer risk among first-degree relatives of TGCT patients and site-specific excess cancer risks in male relatives and in the mothers of TGCT patients. These cancer sites constitute diseases for which there is some prior evidence to suggest a genetic relationship to TGCT. Identification of other cancers as part of the familial TGCT disease spectrum would both provide clinically relevant insight into this syndrome, and enhance the statistical power of gene-seeking linkage analysis.

We propose two studies, each targeting the ITCLC set of high-risk TGCT families, none of which come from the US: (a) Centralized Pathology Review of Familial TGCT; and (b) The Occurrence of Cancer Other than Germ Cell Tumors in TGCT Families. Data will be provided by three of the largest ITCLC contributors; each will contact TGCT probands and their relatives and collect the primary data under their familial and non-familial TGCT, and perform the data analysis for both studies. NCI will neither seek nor receive individual identifying information from any participant. Currently, our UK collaborator has completed acquisition of a Federal Wide Assurance (FWA) and local ethical review. Since this group is contributing 70% of the families in these two projects, we now bring that component before the NCI Special Studies IRB. We shall return to the IRB for review of the other two contributors upon completion of their local ethical review process.

ELIGIBILITY:
* INCLUSION CRITERIA:

The criterion establishing familial TGCT is the presence of at least two cases of documented GCT in blood relatives.

A case will be determined to have TGCT according to the following criteria:

Pathologic confirmation of a germ cell-derived tumor arising in the testis. Estragonadal sperm cell tumors will also be included.

Germ cell-derived histologies including: seminoma, embryonal carcinoma, endodermal sinus (yolk sac) tumor, gonadoblastoma, choriocarcinoma, teratoma, and mixed germ cell tumor.

A case will be determined to have TIN on the basis of pathologic confirmation of intratubular malignant germ cells (ITMGCs) as defined by Burke and Mostofi.

Ages: 4 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families with at least two histopathologically confirmed cases of TGCT, or a combination of TGCT and extragonadal germ cell tumor, and with DNA from at least one affected case will be enrolled at the U.S., U.K., and Norwegian study sites. For the sub-studies, data will be obtained on all family members (siblings, parents, offspring, aunts, uncles, grandparents, cousins) at up to 3 degrees of genetic relatedness to the proband.
Sampling Method: Non-Probability Sample
Enrollment: 1842 (Actual)
Dates: Start 2004-01-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Discovery of new testicular cancer susceptibilitygenes | Duration of Study
  This outcome is the responsibility of the total ITCLC consortium, and will draw upon the collection of DNA samples from multiplecase TGCT families assembled for the purpose of gene discovery. That activity isseparate from the two substudies being proposed in the current document.

SECONDARY OUTCOMES:
Characterization of the familial testicular cancer syndrome phenotype | Duration of Study
  1. We will quantify the risks of cancers (both all sites combined and site-specific risks) other than TGCT in the relatives of multiple-casefamilies. 2. We will perform a central pathology review in which the familial TGCT cases will be compared with age-matched unselected TGCT cases, to determine whether there are unique histologic features which characterize the familial cases.

CONTACTS AND LOCATIONS:
Overall Officials: Mary L McMaster, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mai PL, Friedlander M, Tucker K, Phillips KA, Hogg D, Jewett MA, Lohynska R, Daugaard G, Richard S, Bonaiti-Pellie C, Heidenreich A, Albers P, Bodrogi I, Geczi L, Olah E, Daly PA, Guilford P, Fossa SD, Heimdal K, Liubchenko L, Tjulandin SA, Stoll H, Weber W, Easton DF, Dudakia D, Huddart R, Stratton MR, Einhorn L, Korde L, Nathanson KL, Bishop DT, Rapley EA, Greene MH. The International Testicular Cancer Linkage Consortium: a clinicopathologic descriptive analysis of 461 familial malignant testicular germ cell tumor kindred. Urol Oncol. 2010 Sep-Oct;28(5):492-9. doi: 10.1016/j.urolonc.2008.10.004. Epub 2009 Jan 22. PMID 19162511
- [Background] Nathanson KL, Kanetsky PA, Hawes R, Vaughn DJ, Letrero R, Tucker K, Friedlander M, Phillips KA, Hogg D, Jewett MA, Lohynska R, Daugaard G, Richard S, Chompret A, Bonaiti-Pellie C, Heidenreich A, Olah E, Geczi L, Bodrogi I, Ormiston WJ, Daly PA, Oosterhuis JW, Gillis AJ, Looijenga LH, Guilford P, Fossa SD, Heimdal K, Tjulandin SA, Liubchenko L, Stoll H, Weber W, Rudd M, Huddart R, Crockford GP, Forman D, Oliver DT, Einhorn L, Weber BL, Kramer J, McMaster M, Greene MH, Pike M, Cortessis V, Chen C, Schwartz SM, Bishop DT, Easton DF, Stratton MR, Rapley EA. The Y deletion gr/gr and susceptibility to testicular germ cell tumor. Am J Hum Genet. 2005 Dec;77(6):1034-43. doi: 10.1086/498455. Epub 2005 Oct 24. PMID 16380914
- [Background] Crockford GP, Linger R, Hockley S, Dudakia D, Johnson L, Huddart R, Tucker K, Friedlander M, Phillips KA, Hogg D, Jewett MA, Lohynska R, Daugaard G, Richard S, Chompret A, Bonaiti-Pellie C, Heidenreich A, Albers P, Olah E, Geczi L, Bodrogi I, Ormiston WJ, Daly PA, Guilford P, Fossa SD, Heimdal K, Tjulandin SA, Liubchenko L, Stoll H, Weber W, Forman D, Oliver T, Einhorn L, McMaster M, Kramer J, Greene MH, Weber BL, Nathanson KL, Cortessis V, Easton DF, Bishop DT, Stratton MR, Rapley EA. Genome-wide linkage screen for testicular germ cell tumour susceptibility loci. Hum Mol Genet. 2006 Feb 1;15(3):443-51. doi: 10.1093/hmg/ddi459. Epub 2006 Jan 11. PMID 16407372